CLINICAL TRIAL: NCT06259539
Title: Effectiveness of a YouTube-delivered Nutrition Education Intervention Among Parents of Children With Obesity and Autism: The Intervention Study
Brief Title: A YouTube Curriculum for Children With Autism and Obesity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Woodcock Institute for the Advancement of Neurocognitive Research and Applied Practice (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-FY2023-307
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder; Obesity, Childhood
Keywords: Mixed-methods research; YouTube; Nutrition education
MeSH Terms: conditions — Autism Spectrum Disorder; Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group completed an 8-week virtual, YouTube-delivered nutrition education intervention. They were expected to watch the assigned videos per week at least once and practice the skills and strategies with their child with autism. This group completed all the baseline, mid-point, and end-point data using the questionnaires/surveys on Qualtrics.
  Interventions: Behavioral: YouTube nutrition education
- Control (No Intervention): This group completed all surveys but received no intervention. They received access to all study materials at the end of the study.

INTERVENTIONS:
Behavioral: YouTube nutrition education — For those in the intervention group, the YouTube training modules had step-by-step recipe demonstrations, strategies on how to get your child to eat more new foods, social stories, First-Then visual chart, and other nutrition education materials. All the videos were less than 5 minutes long, and parents were assigned 2 videos per week for 8 consecutive weeks. Parents answered 2 open-ended questions each week related to the educational materials they reviewed.
  Arms: Intervention

SUMMARY:
Parents as primary caregivers play an important role in shaping children's mealtime and eating behaviors; and in preventing weight gain. Conventionally, in-person, parent-implemented treatments have worked well for children with autism, however, post-COVID-19 pandemic there is a need for virtual, evidence-based training for parents to improve nutrition in children with autism and weight issues. This study aims to: a) increase self-efficacy among parents of children with autism and overweight or obesity to feed their children a healthy diet, b) improve parental nutrition knowledge and skills on how to feed their child with autism and overweight or obesity a healthier diet, c) improve their child's mealtime behaviors, and d) increase the child's dietary variety.

DETAILED DESCRIPTION:
This study sought to recruit 24 parents of children with Autism Spectrum Disorder (ASD), and overweight or obesity via emails, digital flyers, and handouts on social media (Facebook), in the USA. This randomized, controlled trial behavioral intervention was conducted from September 2023 to February 2024 and included a YouTube-delivered, 8-week, virtual, nutrition education intervention for the parents.

Participants were randomly allotted to either the intervention or control group by using the randomization (RAND) function on Microsoft Excel. Participants in the intervention group received access to the 16 YouTube videos, educational handbook, recipe modeling, and other training, while participants in the control group only got access to the questionnaires/surveys.

All 8 video modules focused on increasing parental nutrition knowledge, skills, and perceived confidence in making food and nutrition-related decisions to feed their child and address mealtime problems, which aligns with Bandura's Social Cognitive Theory constructs of self-efficacy and behavioral capabilities.

Participants were asked to complete validated questionnaires at baseline, mid-point, and end: parental self-efficacy; the Nutrition knowledge survey; Brief Autism Mealtime Behavior Inventory (BAMBI), followed by a small qualitative open-ended questionnaire for parental feedback on the overall acceptability and satisfaction of the intervention at the end of 8-weeks. All participants were asked to use the ASA-24 (National Cancer Institute) to complete a 24-hour food recall for their child with autism at baseline and end-point.

Demographic data was collected at baseline for all participants. Participants were selected if a) they were 18 years or older; b)had a child with autism between the ages 6 and 11 years c) child's Body Mass Index was > 85th percentile; d) child accepted at least 20 foods e) child did not take any medicines that affect appetite and weight.

ELIGIBILITY:
Inclusion Criteria:

1. Participants have a child between the ages of 6 to 11 years with a diagnosis of autism
2. have a child with autism with a Body Mass Index (BMI) equal to or greater than the 85 percentile
3. they can read and understand English
4. they can access the internet and participate in online research
5. their child with autism accepts at least 20 foods
6. their child with autism is not on a special restricted diet
7. their child with autism does not consume any medications affecting eating.
8. they are 18 years of age or older

Exclusion Criteria:

1. if the child is on medication such as antidepressants, antipsychotics, or SSRIs
2. if the child has high food selectivity (eats less than 20 foods).
3. if the child has a healthy body weight.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-02-10 (Estimated); Study Completion 2024-02-13 (Estimated)

PRIMARY OUTCOMES:
Parental self-efficacy | 8 weeks
  The study utilized a previously validated 9-item list questionnaire that measured their level of confidence (self-efficacy) in their ability to make nutrition-related decisions for their child with autism and overweight or obesity
Parents's nutrition knowledge | 8 weeks
  To test this, a previously validated 18-item questionnaire was administered to test their knowledge of family mealtimes, food groups, and meal planning.

SECONDARY OUTCOMES:
Brief Autism Mealtime Behavior Inventory (BAMBI) | 8 weeks
  This is an 18-item questionnaire designed to evaluate mealtime behaviors in your child with autism.
Child's food intake | 8 weeks
  The Automated Self-Administered 24-hour (ASA24®) dietary assessment tool was used to collect and analyze the child's dietary intake to monitor any changes pre and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Miteshri D Prajapati, M.S, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Denton, Texas, United States